CLINICAL TRIAL: NCT02905123
Title: Brief Internet Intervention for Hazardous Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 075/2016
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Check Your Drinking (CYD) (Experimental): The CYD is a brief online intervention designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Interventions: Behavioral: Check Your Drinking
- Control (No Intervention): No Intervention Control

INTERVENTIONS:
Behavioral: Check Your Drinking
  Arms: Check Your Drinking (CYD)

SUMMARY:
Amazon's Mechanical Turk (MTurk) is an online platform that has become a popular means of recruiting participants with problem drinking, gambling, or even illicit drug use for the purposes of survey-based research. There is also the possibility that potential participants could be identified through MTurk for online longitudinal studies, including for brief intervention research. The potential to quickly and easily identify large numbers of participants through MTurk is important for research evaluating online interventions during the period that these interventions are being developed and refined. However, before proposing MTurk workers as a viable source for participants in online intervention trials, it is important to evaluate the feasibility of using MTurk for such a purpose. This pilot study proposes to test this feasibility by systematically replicating a trial of an extensively evaluated brief online intervention for hazardous alcohol use (CheckYourDrinking; CYD) and will attempt to recruit and follow-up participants for this replication using people recruited through MTurk.

Participants will be recruited through Amazon's MTurk crowdsourcing platform. Participants identified as problem drinkers based on an initial survey will be invited to complete another survey in 3 months time. Those who are interested will be randomized to receive access to the Check Your Drinking screener (CYD condition) or to a no additional information condition (control condition). At three-months post-baseline, the MTurk portal will be used to send invitation emails that contain a link to the follow-up survey. The primary hypothesis to be tested is that participants receiving access to the CYD intervention will report a greater level of reduction in number of drinks in a typical week between the baseline survey and three-month follow-up as compared to participants in the no information control condition.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Use Disorders Identification Test (AUDIT) score of 8 or more
* Willingness to complete a 3-month follow-up survey
* 18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of drinks consumed during a typical week | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No